CLINICAL TRIAL: NCT03551366
Title: Efficacy of Skill Acquisition Methods Underpinning Pedagogy for LEarning in Physical Education (SAMPLE-PE) in Children Aged 5-6 Years
Brief Title: Influence of Different Physical Education Pedagogical Approaches on the Health and Development of 5-6 Year Old Children
Acronym: SAMPLE-PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Universität Münster (Other); University of Strathclyde (Other); University of Otago (Other); Victoria University (Unknown); Newcastle University (Other); University of Rome Foro Italico (Other)
Responsible Party: Principal Investigator, James Rudd, Senior Lecturer In Physical Education, Liverpool John Moores University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LiverpoolJMU
Record Dates: First submitted 2018-05-10; First posted 2018-06-11 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Child; Child Development; Health Behavior; Physical Activity
Keywords: Physical Activity; Physical Education; Children; Pedagogy; Motor Competence; Perceived Motor Competence; Self-perception; Cognition; Fundamental Movement Skills
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Schools are randomly assigned to either a control (usual practice), linear PE pedagogy or nonlinear PE pedagogy arm. Both linear and nonlinear arms will receive 15 weeks of physical education lessons from trained coaches, whereas the control group will carry on with PE lessons as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Subjects in this group will continue with their usual PE curriculum for 15 weeks.
- Linear (Experimental): Subjects in this group will receive a linear PE curriculum for 15 weeks. Linear Pedagogy is underpinned by neuro-computation approach to motor learning such as information processing theory and prescribes that an ideal movement pattern exists for each task and that the teacher's role is to help learners recreate that pattern. Furthermore, theorists have suggested that learning is a gradual, linear process. This linear pedagogy is supported by a teaching and learning approach that includes both prescriptive and repetitive actions, utilising technical demonstrations that provide learners with a 'visual template or criterion model' for the desired skill . As a consequence, a PE pedagogy has developed whereby the teacher's role is to make all the decisions, and the learner's role is to follow their instructions on cue - a teacher-led approach to PE.
  Interventions: Behavioral: Linear
- Nonlinear (Experimental): Subjects in this group will receive a nonlinear PE curriculum for 15 weeks. Nonlinear pedagogy is grounded in Ecological Dynamics theory. Ecological dynamics regards learners as complex adaptive systems which afford opportunities for action from their environment and generate movement solutions to satisfy the combination of personal, environmental and task constraints imposed upon them. According to nonlinear pedagogy, the teacher's role is to design learning experiences that create behavioural symmetry between learning and the performance environment. The teacher is a facilitator and manipulates constraints to channel the learner's physical development, while learners are left free to experiment and select the movement solutions that best answer their individual needs. This child-focused, less prescriptive approach may enhance a child's intrinsic motivation by offering freedom to choose, and an emphasis on exploration and problem solving.
  Interventions: Behavioral: Nonlinear

INTERVENTIONS:
Behavioral: Linear — The linear pedagogy arms consists of three, five-week phases of lesson delivery, commencing around two weeks after baseline assessments. The first phase focuses on dance, the second on gymnastics and the final phase on ball sports. Each phase has its own schemes of work which includes five lessons objectives, each taught over a two lesson period. The lesson objectives aligned to the aims of English national curriculum. Lessons are delivered twice a week by trained coaches, with each lesson lasting 60 minutes in total, with 45 minutes of on task teaching time. Linear curriculum lessons will be focused on the functioning of the body and children learning movement patterns. These lessons will be far more prescriptive and have clearly stated outcomes/goals for each lesson, with a typical lesson structure following the structure of warm up, isolated practice of technique or skill, simulated game and warm down.
  Arms: Linear
Behavioral: Nonlinear — The non-linear pedagogy arm consists of three, five-week phases of lesson delivery, commencing around two weeks after baseline assessments. The first phase focuses on dance, the second on gymnastics and the final phase on ball sports. Each phase has its own schemes of work which includes five lessons objectives, each taught over a two lesson period. The lesson objectives align to the aims of English national curriculum. Lessons are delivered twice a week by trained coaches, with each lesson lasting 60 minutes in total, with 45 minutes of on task teaching time. The nonlinear curriculum lessons will look to make sure that children are both engaged and empowered throughout the learning process. In adherence to representative learning design, we will look to contextualise lessons and guide learning through the use of books/stories, lived experiences and the sharing of ideas.
  Arms: Nonlinear

SUMMARY:
The Skill Acquisition Methods underpinning Pedagogy for LEarning in Physical Education (SAMPLE-PE) project aims to investigate the influence of different pedagogical approaches to teaching and learning in physical education (PE) on 5-6 year old children's health and development. Schools from deprived areas are invited to take part in the project and will be randomly assigned to either: (1) linear pedagogy PE curriculum programme, (2) nonlinear pedagogy PE curriculum programme or (3) carry on as normal. The linear and nonlinear pedagogy PE programmes will be underpinned by different and contrasting theories of skill acquisition and are delivered by trained coaches over 15 weeks. Children will be measured to assess their physical, psychological, cognitive, and emotional health and development, and their physical activity levels at the start of the study, immediately after the 15 week PE programme, and again after 12 months. It is expected that children taking part in the linear and nonlinear PE programmes will demonstrate greater physical development than children attending schools that carry on as normal. Furthermore, it is also anticipated that children taking part in the nonlinear PE programme will show greater gains in psychological, cognitive and emotional outcomes than the linear and usual practice programmes.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-6 years attending Liverpool primary schools.

Exclusion Criteria:

* From the details given in participant's Child Medical Form, any child diagnosed with health or co-ordination issues that could affect motor competency will be excluded from analyses.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 361 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline motor competence level (Locomotor and Object-Control Skills) at 5 and 12 months | Baseline (month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Fundamental motor skill competency in locomotor and object control skills will be assessed using the Test of Gross Motor Development-3 (TGMD-3: Ulrich, 2013; Webster and Ulrich, 2017).
Change from baseline stability skill level at 5 and 12 months | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Fundamental motor skill competency in stability category skills will be assessed using the Test of Stability skills (Rudd et al., 2015).
Change from baseline motor creativity level at 5 and 12 months | Baseline (month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Motor creativity will be assessed using the Divergent Movement Ability Assessment (Cleland and Gallahue, 1993)

SECONDARY OUTCOMES:
Change from Baseline Physical Activity at 5 and 12 Months | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Physical Activity will be assessed by wrist-worn accelerometers (ActiGraph GT9X+) on their non-dominant wrist continuously for seven days. Parents are asked to keep a diary on when the monitor was has been worn.
Change from Baseline Perceived Physical Competence at 5 and 12 Months | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Perceived Physical competence will be assessed using the corresponding subscale within The Pictorial Scale of Perceived Competence and Social Acceptance for Young Children (Harter & Pike, 1984). The Physical Competence subscale includes items 3, 7, 11, 15, 19, and 23 from the Pictorial Scale. Each item is scored on a 4-point scale, where 4 represents the highest degree of perceived competence. The subscale score is computed by adding values of child responses and ranges from 6 to 24.
Change from Baseline Perceived Movement Skill Competence at 5 and 12 Months | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Perceived Skill Competence will be assessed by the Pictorial Scale of Perceived Movement Skill Competence for Young Children (Barnett et al., 2015).
  The Scale consists of twelve items with two subscales of six items each representing "Locomotor Skill Perceived Competence" and "Object-Control Skill Perceived Competence", respectively. Each item is scored on a 4-point scale, where 4 represents the highest degree of perceived competence. Subscale scores are computed by adding values of child responses and range from 6 to 24 (higher values indicate higher perceived competence).
  All 12 items are summed to generate the Perceived Movement Skill Competence scale score, which ranges from 12 to 48 (higher values indicate higher perceived competence).
Change from Baseline Motivation at 5 months | Baseline (Month 0) and after the intervention (approximately 5 months post-baseline)
  Self Determined Motivation in children will be assessed by a write, draw, show and tell, method, adapted from Noonan et al. (2017).
Change from Baseline Executive Functions at 5 and 12 Months | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Executive functions will be assessed by three activities from the National Institute for Health toolbox (Weintraub et al., 2013; Zelazo & Bauer, 2013)
Change from Baseline Self-Regulation at 5 and 12 Months (Strengths and Difficulties Questionnaire) | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Self-Regulation will be assessed by the Strength and Difficulties Questionnaire (Goodman, 1997; Stone et al., 2010), as completed by the child's class teacher.
  The Strength and Difficulties Questionnaire consists of 25 items within 5 subscales (emotional, conduct, hyperactivity, peer and prosocial).
  There are five items on each subscale with each item scored 0, 1 or 2. Scores therefore range from 0-10 for each subscale, with 10 indicating higher levels of difficulties (emotional, conduct, hyperactivity, peer subscales) or strengths (prosocial subscale) and 0 indicating lower levels.
  A total difficulties score is also generated by summing scores from all the scales except the prosocial scale, with scores ranging from 0 (low) to 40 (high).
Change from Baseline Self-Regulation at 5 and 12 Months (Response to Challenge Scale) | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Self-Regulation will be assessed by the Response to Challenge Scale (RCS: Lakes, 2012; 2013)
  The RCS is an observer-rated measure of children's responses to a physical challenge and includes 16 bipolar adjectives (e.g., Vulnerable-Invincible) rated on 7-point scales (scored 1-7).
  There are three subscales assessed: "Cognitive" (6 items, scoring range from 6 to 42), "Affective" (7 items, scoring range from 7 to 49) and "Physical/Motor" (3 items, scoring range from 3 to 21). Negatively worded items are reversed prior to aggregation, so that possible scores on all subscales ranged from 1 to 7, with higher scores indicating greater self-regulation.
Body Mass Index | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Stature (to the nearest 0.1cm) and mass (to the nearest 0.1kg) will be assessed to calculate and report BMI in kg/m^2
Maturation | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Stature, mass, and sitting height will be combined to determine maturation status using an age and sex specific maturity offset calculation (Mirwald et al., 2002).
Waist girth | Baseline (Month 0), after the intervention (approximately 5 months post-baseline) and follow-up (approximately 12 month post-baseline)
  Waist girth (nearest 0.1cm) will be assessed as marker of central adiposity

CONTACTS AND LOCATIONS:
Overall Officials: James Rudd, PhD, Principal Investigator — Liverpool John Moores
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee MC, Chow JY, Komar J, Tan CW, Button C. Nonlinear pedagogy: an effective approach to cater for individual differences in learning a sports skill. PLoS One. 2014 Aug 20;9(8):e104744. doi: 10.1371/journal.pone.0104744. eCollection 2014. PMID 25140822
- [Background] Tompsett C, Sanders R, Taylor C, Cobley S. Pedagogical Approaches to and Effects of Fundamental Movement Skill Interventions on Health Outcomes: A Systematic Review. Sports Med. 2017 Sep;47(9):1795-1819. doi: 10.1007/s40279-017-0697-z. PMID 28213755
- [Background] Chow JY, Davids K, Button C, Shuttleworth R, Renshaw I, Araujo D. Nonlinear pedagogy: a constraints-led framework for understanding emergence of game play and movement skills. Nonlinear Dynamics Psychol Life Sci. 2006 Jan;10(1):71-103. PMID 16393504
- [Background] Rudd JR, Barnett LM, Butson ML, Farrow D, Berry J, Polman RC. Fundamental Movement Skills Are More than Run, Throw and Catch: The Role of Stability Skills. PLoS One. 2015 Oct 15;10(10):e0140224. doi: 10.1371/journal.pone.0140224. eCollection 2015. PMID 26468644
- [Background] Ulrich DA, The test of gross motor development-3 (TGMD-3): Administration, scoring, and international norms. Spor Bilimleri Dergisi 24(2): 27-33, 2013.
- [Background] Cleland FE, Gallahue DL. Young children's divergent movement ability. Percept Mot Skills. 1993 Oct;77(2):535-44. doi: 10.2466/pms.1993.77.2.535. PMID 8247678
- [Background] Barnett LM, Ridgers ND, Zask A, Salmon J. Face validity and reliability of a pictorial instrument for assessing fundamental movement skill perceived competence in young children. J Sci Med Sport. 2015 Jan;18(1):98-102. doi: 10.1016/j.jsams.2013.12.004. Epub 2014 Jan 2. PMID 24485803
- [Background] Barnett LM, Robinson LE, Webster EK, Ridgers ND. Reliability of the Pictorial Scale of Perceived Movement Skill Competence in 2 Diverse Samples of Young Children. J Phys Act Health. 2015 Aug;12(8):1045-51. doi: 10.1123/jpah.2014-0141. Epub 2014 Sep 22. PMID 25243542
- [Background] Noonan RJ, Fairclough SJ, Knowles ZR, Boddy LM. One Size Does Not Fit All: Contextualising Family Physical Activity Using a Write, Draw, Show and Tell Approach. Children (Basel). 2017 Jul 14;4(7):59. doi: 10.3390/children4070059. PMID 28708114
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Harter S, Pike R. The pictorial scale of perceived competence and social acceptance for young children. Child Dev. 1984 Dec;55(6):1969-82. PMID 6525886
- [Background] Weintraub S, Dikmen SS, Heaton RK, Tulsky DS, Zelazo PD, Bauer PJ, Carlozzi NE, Slotkin J, Blitz D, Wallner-Allen K, Fox NA, Beaumont JL, Mungas D, Nowinski CJ, Richler J, Deocampo JA, Anderson JE, Manly JJ, Borosh B, Havlik R, Conway K, Edwards E, Freund L, King JW, Moy C, Witt E, Gershon RC. Cognition assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S54-64. doi: 10.1212/WNL.0b013e3182872ded. PMID 23479546
- [Background] Fox NA. Commentary on Zelazo and Bauer (editors), National Institutes of Health Toolbox Cognition Battery (CB): validation for children between 3 and 15 years. Monogr Soc Res Child Dev. 2013 Aug;78(4):150-5. doi: 10.1111/mono.12044. No abstract available. PMID 23952209
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Stone LL, Otten R, Engels RC, Vermulst AA, Janssens JM. Psychometric properties of the parent and teacher versions of the strengths and difficulties questionnaire for 4- to 12-year-olds: a review. Clin Child Fam Psychol Rev. 2010 Sep;13(3):254-74. doi: 10.1007/s10567-010-0071-2. PMID 20589428
- [Background] Lakes KD. The Response to Challenge Scale (RCS): The Development and Construct Validity of an Observer-Rated Measure of Children's Self-Regulation. Int J Educ Psychol Assess. 2012 Apr;10(1):83-96. PMID 25750758
- [Background] Lakes KD. Measuring self-regulation in a physically active context: Psychometric analyses of scores derived from an observer-rated measure of self-regulation. Ment Health Phys Act. 2013 Oct;8(3):189-196. doi: 10.1016/j.mhpa.2013.09.003. PMID 25750662
- [Background] Mirwald RL, Baxter-Jones AD, Bailey DA, Beunen GP. An assessment of maturity from anthropometric measurements. Med Sci Sports Exerc. 2002 Apr;34(4):689-94. doi: 10.1097/00005768-200204000-00020. PMID 11932580
- [Derived] Rudd JR, Crotti M, Fitton-Davies K, O'Callaghan L, Bardid F, Utesch T, Roberts S, Boddy LM, Cronin CJ, Knowles Z, Foulkes J, Watson PM, Pesce C, Button C, Lubans DR, Buszard T, Walsh B, Foweather L. Skill Acquisition Methods Fostering Physical Literacy in Early-Physical Education (SAMPLE-PE): Rationale and Study Protocol for a Cluster Randomized Controlled Trial in 5-6-Year-Old Children From Deprived Areas of North West England. Front Psychol. 2020 Jun 17;11:1228. doi: 10.3389/fpsyg.2020.01228. eCollection 2020. PMID 32625143